CLINICAL TRIAL: NCT00961610
Title: Internet-based Support in the Rehabilitation of Danish Cancer Survivors
Brief Title: Internet-based Support in Cancer Rehabilitation
Status: Completed | Type: Observational
Sponsor: Danish Cancer Society (Other)
Collaborators: TrygFonden, Denmark (Industry); IMK Almene Fond (Other)
Responsible Party: Christoffer Johansen, Department of Psychosocial Cancer Research
Other Study IDs: PP-07024
Record Dates: First submitted 2009-08-17; First posted 2009-08-19 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Cancer
Keywords: internet support; cancer; rehabilitation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Internet support group Intervention
  Interventions: Behavioral: Internet peer-support group
- Control group
  Interventions: Behavioral: Internet peer-support group

INTERVENTIONS:
Behavioral: Internet peer-support group — The Internet peer-support groups provided a self-guided space for communication, including an Internet discussion forum, a live chat room and a personal message system. No therapeutic content or information services were offered within the groups.
  All Internet groups were run in a browser-based software platform with access through the website of the Danish Cancer Society (http://www.cancer.dk). All discussions were protected by a password and communication was encrypted.
  The Internet groups in this study were all closed peer-support groups, accessible only by an invitation received by e-mail after registration for the study. The groups were open to access 24 h a day for 13 months from their individual starting date.

SUMMARY:
This 2-arm randomized trial assessed the incremental effect of providing a lecture on Internet use followed by participation in an Internet-based peer support group following a week-long rehabilitation program, over and above any possible general effect of participation in the rehabilitation program.

Primary outcome measures are adjustment to cancer and mood disturbance.

ELIGIBILITY:
Inclusion Criteria:

* Cancer survivors who were randomized for or self-selected to a rehabilitation course at the Dallund Rehabilitation Centre were included in the study.

Exclusion Criteria:

* Rehabilitation course weeks in which cancer survivors over 50 years of age were targeted specifically were excluded.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 66 scheduled rehabilitation course weeks were screened for eligibility between 19 April 2004 and 31 December 2005 from the Rehabilitation Centre Dallund in Denmark. All 58 eligible courses including 921 individuals were enrolled and randomized as 27 case weeks (n = 416 persons) and 31 control weeks (n = 505 persons). Baseline assessments were obtained from 799 individuals. Data from 10 individuals (5 from each treatment group) were subsequently excluded, as they did not attend a rehabilitation course week as planned, leaving final study population of 794 individuals analyzed by 'intention-to-treat' (case: n = 361/794; control: n = 433/794). Participants were followed up for 12 months in accordance with their dates of attendance of the rehabilitation course from 19 April 2004 till 31 December 2006.
Sampling Method: Probability Sample
Enrollment: 794 (Actual)
Dates: Start 2004-04; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Adjustment to cancer measured by the Mini-MAC scale Mood disturbance measured by POMS-SF scale

SECONDARY OUTCOMES:
Self-rated global health

CONTACTS AND LOCATIONS:
Overall Officials: Christoffer Johansen, MD, PhD, DrMedSci, Principal Investigator — Department of Psychosocial Cancer Research
Locations (1):
- Department of Psychsocial Cancer Research, Copenhagen, Denmark